CLINICAL TRIAL: NCT04439565
Title: Study on Susceptibility Genes and Pathogenic Mechanism of Non-syndromic Familial Aortic Dissection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Medical Association (Network)
Responsible Party: Principal Investigator, Zaiping Jing, professor, Chinese Medical Association
Other Study IDs: https://orcid.org/0000-0002-05
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Aortic Dissection; Family Research; Aortic Dissection, Familial, With or Without Aortic Aneurysm
Keywords: aortic dissection; pathogenesis; familial inheritance; susceptibility gene
MeSH Terms: conditions — Aortic Dissection | interventions — Movement

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA is extracted from blood and preserved for a long time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: movement — aortic dissection or aneurysm patients this is an observation cohort study about a Non-syndromic Familial Aortic Dissection without intervention.

SUMMARY:
Aortic dissection is dangerous and difficult to predict, so it is particularly important to carry out early prevention, diagnosis and rational treatment for high-risk groups. The related genes found in previous studies can not be detected in all patients with dissection; at present, the pathogenesis of non-syndromic aortic dissection is not clear, of which about 20% of patients have family aggregation and have the general representative characteristics of non-syndromic dissection. In this project, the peripheral blood samples of core family subjects were detected by sequencing technique. analyze disease-related susceptibility genes; 2 determine the effect of susceptibility genes on the incidence of dissection in mice through animal experiments; and 3 explore the effect of susceptibility genes on cell function at the cellular level.

ELIGIBILITY:
Inclusion Criteria:

* Family inclusion criteria: 1 at least one person in each generation of a family has aortic dissection, and at least two generations of members can be included;

Exclusion Criteria:

* Pedigree exclusion criteria: pedigree members have marfan syndrome, Loeys-Dietz syndrome, Ehler-Danlos syndrome, aneurysm-Osteoarthritis syndrome and other syndroms

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1, family members have no traumatic aortic dissection; 2, no pregnancy or tumor.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-17 (Estimated); Primary Completion 2023-06-17 (Estimated); Study Completion 2023-07-17 (Estimated)

PRIMARY OUTCOMES:
gege | 2023
  Discovery of known or unknown genes

CONTACTS AND LOCATIONS:
Locations (1):
- Changhaihospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided